CLINICAL TRIAL: NCT05401032
Title: TryptoBPH - Proof-of-concept Study to Evaluate the Safety and Efficacy of Tryptophan in Patients with BPH
Brief Title: Proof-of-concept Study to Evaluate the Safety and Efficacy of Tryptophan in Patients with BPH.
Acronym: TryptoBPH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Clinical Academic Center (2CA-Braga) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TryptoBPH; 2024-519076-75-00 (EU CTIS Number); 2021-000946-16 (EudraCT Number)
Record Dates: First submitted 2022-05-25; First posted 2022-06-02 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: BPH; LUTS(Lower Urinary Tract Symptoms)
Keywords: BPH; LUTS; 5-HTP; Oxitriptan; Tamsulosin
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: Single-center, parallel group, randomized clinical trial designed to evaluate the effect of treatment with 5-HTP, comparative to Tamsulosin, for a period of 6 months, on LUTS, changes in urine maximum flow rate (Qmax), prostate volume, erectile function and quality of life due to urinary symptoms in adult patients with BPH.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Complete (double) blinding is not possible to achieve, nonetheless, in order to lessen assessment bias, efficacy and safety assessment procedures will be performed by the assigned blinded research staff. In order to assure blinding across the study, randomization data will be kept confidential and will not be accessible to anyone, except to unblinded research staff, pharmacy staff. Both groups will be monitored for the same study duration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm (Active Comparator): tamsulosin 0.4mg (once a day) for 6 months.
  Interventions: Drug: Tamsulosin
- Experimental arm (Experimental): 5-hidroxitriptophan 100 mg (3 times a day) for 6 months.
  Interventions: Drug: 5-hidroxitriptophan

INTERVENTIONS:
Drug: Tamsulosin — Oral medication, once a day for 6 months.
  Other Names: Omnic
  Arms: Control arm
Drug: 5-hidroxitriptophan — Oral medication, 3 times a day for 6 months.
  Other Names: Cincofarm
  Arms: Experimental arm

SUMMARY:
Benign prostatic hyperplasia (BPH) is one of the most prevalent human diseases and a major cause of lower urinary tract symptoms (LUTS). Some men respond to current medical treatment (mainly α-1 adrenoreceptor antagonists and 5 α-reductase inhibitors), but a large proportion of patients continues to need a surgical procedure to treat resistant LUTS or even more serious complications of BPH, creating the emerging necessity for novel pharmacological therapies.

Oxitriptan may have a possible positive effect on BPH associated symptoms with probably no impact in sexual function (which is a common side effect of the current drugs for BPH associated symptoms). Also, improvement in symptoms could be higher than that of current drugs used for this condition.

This is a single-center parallel group, randomized clinical trial. The study will take place in Hospital de Braga (Urology department). Eligible patients will be randomized to receive tamsulosin 0.4mg (once a day, q.d.) or 5-HTP (5-hidroxitriptophan) 100mg (three times a day, t.i.d.), for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* Male patients with BPH for which tamsulosin is the therapeutic option per SoC;
* Aged ≥50 and less than 75 years old;
* With prostate volume ≥30 cm3 by TRUS;
* Diagnosed with LUTS defined by a stable IPSS total score ≥13 points.

Exclusion Criteria:

* Patients with post-void bladder residual volume ≥250 ml;
* Patients with intravesical obstruction from any cause other than BPH;
* History of any procedure considered an intervention for BPH;
* Patients with active urinary tract infection;
* History of recurrent urinary tract infections;
* Current prostatitis or diagnosis of chronic prostatitis;
* History of prostate or invasive bladder cancer;
* Use of 5 α-reductase inhibitors within 6 months;
* Phytotherapy within 2 weeks before entry;
* Use of serotonin reuptake inhibitors or monoamine oxidase inhibitors;
* Patients with acute or chronic kidney failure;
* Patients with diagnosed or suspicion of intolerance to lactose;
* Patients submitted to general anesthesia in the past 4 weeks;
* Known intellectual disability that may hampers giving informed consent and would make the patient inappropriate for entry into this study, in the judgment of the investigator.

Ages: 50 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) | Change from baseline to day 1, 1-month, 3- month and EOT (6-month)
  Evaluate the effect of tryptophan supplementation on lower urinary tract symptoms (LUTS)

SECONDARY OUTCOMES:
Qmax | Change from baseline to EOT (6-month)
  Urine maximum flow rate
IIEF-5 | Change from baseline to EOT (6-month)
  Erectile function, assessed by International Index of Erectile Function-5 (IIEF-5)
Prostate volume | Change from baseline to EOT (6-month)
  Prostate volume (in cc), assessed by trans-rectal ultra-sound
question 8 of the IPSS | Change from baseline to EOT (6-month)
  quality of life due to urinary symptoms (question 8 of the IPSS).

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Dias, Principal Investigator — Hospital de Braga
Locations (1):
- Clinical Academic Center - Braga, Association (2CA-Braga), Braga, Portugal

IPD SHARING:
Plan to Share IPD: Undecided